CLINICAL TRIAL: NCT02986516
Title: Title of Study: SAcral Chordoma: a Randomized & Observational Study on Surgery Versus Definitive Radiation Therapy in Primary Localized Disease (SACRO)
Brief Title: Sacral Chordoma: Surgery Versus Definitive Radiation Therapy in Primary Localized Disease
Acronym: SACRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Italian Sarcoma Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISG SACRO
Record Dates: First submitted 2016-12-02; First posted 2016-12-08 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Chordoma
MeSH Terms: conditions — Chordoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomized Cohort (Experimental): Participants who will decided to undergo to randomization, will receive surgical treatment or definitive radiotherapy according with randomization assignment
  Interventions: Other: Randomized Cohort
- Prospective Cohort (Active Comparator): Participants who will not decide to be randomized, will received the surgical or definite radiotherapy treatment according to their choice
  Interventions: Radiation: Prospective cohort

INTERVENTIONS:
Other: Randomized Cohort — Surgical treatment with different approach, based on the characteristics of the tumor or definitive high dose radiotherapy (carbon ion radiotherapy, proton-therapy, mixed photons-proton therapy) will be assigned by randomization
  Arms: Randomized Cohort
Radiation: Prospective cohort — Surgical treatment or definitive high dose radiotherapy will be selected by the patients and will be prospectively evaluated
  Arms: Prospective Cohort

SUMMARY:
Comparative study on surgery versus definitive radiation therapy in primary localized sacral chordoma

DETAILED DESCRIPTION:
International, multicenter, comparative, open-label, parallel-group, mixed Observational-Randomized Controlled Trial.

All the patients, who are candidate for the study will receive full information on the characteristics, potential effectiveness and side effects of the two alternatives treatments: radiotherapy (RT) and surgical treatment Eligible patients will be asked to be randomized in order to receive treatment A (surgery, with or without RT) or treatment B (definitive RT) Who will refuse randomization will be included in the Prospective Cohort Study (PCS) and will be treated accordingly to their choice (treatment option A or treatment option B).

The same radiotherapy and surgical regimen will be administered in the PCS and in the Randomized Clinical Trial (RCT) cohort

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis (brachyury expression) of primary sacral chordoma,of any diameter and arising at any site from S1 to coccyx.
* Age≥18years
* ECOG-performance status (PS) 0-2
* No previous antineoplastic therapy
* Macroscopic tumor detectable at MRI/CT scan
* Patient amenable for surgery
* Patient amenable for RT
* Written informed consent given before the enrolment, according to International Conference on Harmonisation/good clinical practice (ICH/GCP).

Exclusion Criteria:

* Distant metastasis
* Inability to maintain treatment position
* Prior radiotherapy to the pelvic region
* Prior therapy for sacral chordoma (including surgery, cryoablation, hyperthermia, etc)
* Local conditions that increase the risk of RT toxicity (tumor ulcerated skin infiltration, non-healing soft tissue infection, fistula in treatment field)
* Rectal wall infiltration
* General conditions that increase the risk of RT toxicity (active sclerodermia, xeroderma pigmentosum, cutaneous porphyria)
* Presence of a second active cancer (with the exception of non-melanoma skin cancer in-situ cervix neoplasia and other in-situ neoplasia)
* Severe comorbidities resulting in a prognosis of less than 6 months
* Inability to give informed consent
* Other malignancy within the last 5 years
* Performance status ≥ 2 (ECOG).
* Significant cardiovascular disease (for example, dyspnea > 2 NYHA)
* Significant systemic diseases grade >3 on the NCI-CTCAE v4.03 scale, that limit patient availability, or according to investigator judgment may contribute significantly to treatment toxicity
* Women who are pregnant or breast-feeding
* Psychological, familial, social or geographic circumstances that limit the patient's ability to comply with the protocol or informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Relapse Free Survival (RFS) | 5 years
  The time from randomization or treatment start date to the date of local disease relapse, distant disease relapse, second primary malignancy or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival (OS) | The patients will be followed in term of Overall Survival, for all the study period (expected average: 10 years)
  The time from randomization or treatment start date to the date of death from any cause
Survival Post Progression (SPP) | Expected average: 36 months
  The time from local disease relapse, distant disease relapse or second primary malignancy, whichever occurred first, to the date of death from any cause
Local Relapse Failure (LRF) | Expected average: 60 months
  The time from randomization or treatment start date to the date of local disease relapse
Distant Relapse Failure (DRF) | Expected average: 60 months
  The time from randomization or treatment start date to the date of distant disease relapse
Best Response rate to definitive radiotherapy | At 12 months, 2 years and 5 years after radiotherapy
  Best Response rate to definitive radiotherapy
Time to best response rate to definitive radiotherapy | At 12 months, 2 years and 5 years after radiotherapy
  Time to best response rate to definitive radiotherapy
Adverse Events Incidence | At end of treatment , 6 months , 12 months 2 years and 5 years after surgery or radiotherapy
  Adverse Events incidence
Evaluation of quality of life measured with Functional Assessment of Cancer Therapy General | every 6 months (expected average: 5 years)
  Evaluation of quality of life measured with Functional Assessment of Cancer Therapy General
Evaluation of quality of life measured with Brief Inventory Pain questionnaires | every 6 months (expected average: 5 years)
  Evaluation of quality of life measured with Brief Inventory Pain questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Gronchi, MD, Principal Investigator — Istituto Nazionale Tumori Milan-Italy; Piero Fossati, MD, Principal Investigator — MedAustron Graz-Austria
Locations (28):
- Austria (2):
  - Medical University of Graz, Graz
  - EBG GmbH MedAustron, Wiener Neustadt, Österreich
- Germany (4):
  - Medical Faculty Carl Gustav Carus Faculty of Medicine, Department of Radiation Oncology,, Dresden
  - University Hospital Carl Gustav Carus Dresden, Dresden
  - University Hospital Essen. West German Proton Therapy Center Essen, Essen
  - Heidelberg Ion-Beam Therapy Center - HIT, Heidelberg
- National Center for Spinal Disorders, Budapest, Hungary
- Italy (9):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI
  - Istituto Ortopedico Rizzoli, Bologna
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Istituto Clinico Humanitas, Milan
  - I.R.C.C.S. Istituto Ortopedico Galeazzi, Milan
  - Centro Nazionale di Adroterapia Oncologica - CNAO, Pavia
  - II Clinica Universitaria Ortopedia e Traumatologia AO Pisa, Pisa
  - Istituto Regina Elena - IFO, Rome
  - Agenzia Provinciale per la Protonterapia - AtreP, Trento
- Saitama Medical Center, Saitama, Japan
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - Leiden University Medical Center, Leiden
- Norwegian Radium Hospital/Oslo Univeristi Hospital, Oslo, Norway
- Centrum Onkologii-Instytut im. Marii Skłodowskiej-Curie, Warsaw, Poland
- Spain (5):
  - H. Val D'Hebron, Barcelona
  - Hosptial San Pau, Barcelona
  - H. San Carlos, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Doctor Peset, Valencia
- United Kingdom (2):
  - The Royal Orthopaedic Hospital, Birmingham
  - Royal National Orthopaedic Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stiller CA, Trama A, Brewster DH, Verne J, Bouchardy C, Navarro C, Chirlaque MD, Marcos-Gragera R, Visser O, Serraino D, Weiderpass E, Dei Tos AP, Ascoli V; RARECARE Working Group. Descriptive epidemiology of Kaposi sarcoma in Europe. Report from the RARECARE project. Cancer Epidemiol. 2014 Dec;38(6):670-8. doi: 10.1016/j.canep.2014.09.009. Epub 2014 Oct 22. PMID 25454979
- [Background] Tirabosco R, Mangham DC, Rosenberg AE, Vujovic S, Bousdras K, Pizzolitto S, De Maglio G, den Bakker MA, Di Francesco L, Kalil RK, Athanasou NA, O'Donnell P, McCarthy EF, Flanagan AM. Brachyury expression in extra-axial skeletal and soft tissue chordomas: a marker that distinguishes chordoma from mixed tumor/myoepithelioma/parachordoma in soft tissue. Am J Surg Pathol. 2008 Apr;32(4):572-80. doi: 10.1097/PAS.0b013e31815b693a. PMID 18301055
- [Background] Brien EW, Mirra JM, Ippolito V. Chondroblastoma arising from a nonepiphyseal site. Skeletal Radiol. 1995 Apr;24(3):220-2. doi: 10.1007/BF00228930. PMID 7610417
- [Background] Vujovic S, Henderson S, Presneau N, Odell E, Jacques TS, Tirabosco R, Boshoff C, Flanagan AM. Brachyury, a crucial regulator of notochordal development, is a novel biomarker for chordomas. J Pathol. 2006 Jun;209(2):157-65. doi: 10.1002/path.1969. PMID 16538613
- [Background] Miozzo M, Dalpra L, Riva P, Volonta M, Macciardi F, Pericotti S, Tibiletti MG, Cerati M, Rohde K, Larizza L, Fuhrman Conti AM. A tumor suppressor locus in familial and sporadic chordoma maps to 1p36. Int J Cancer. 2000 Jul 1;87(1):68-72. PMID 10861454
- [Background] Kelley MJ, Korczak JF, Sheridan E, Yang X, Goldstein AM, Parry DM. Familial chordoma, a tumor of notochordal remnants, is linked to chromosome 7q33. Am J Hum Genet. 2001 Aug;69(2):454-60. doi: 10.1086/321982. Epub 2001 Jul 10. PMID 11452362
- [Background] Lee-Jones L, Aligianis I, Davies PA, Puga A, Farndon PA, Stemmer-Rachamimov A, Ramesh V, Sampson JR. Sacrococcygeal chordomas in patients with tuberous sclerosis complex show somatic loss of TSC1 or TSC2. Genes Chromosomes Cancer. 2004 Sep;41(1):80-5. doi: 10.1002/gcc.20052. PMID 15236319
- [Background] Dutton RV, Singleton EB. Tuberous sclerosis: a case report with aortic aneurysm and unusual rib changes. Pediatr Radiol. 1975 Jun 13;3(3):184-6. doi: 10.1007/BF01006909. PMID 1233436
- [Background] Yang XR, Ng D, Alcorta DA, Liebsch NJ, Sheridan E, Li S, Goldstein AM, Parry DM, Kelley MJ. T (brachyury) gene duplication confers major susceptibility to familial chordoma. Nat Genet. 2009 Nov;41(11):1176-8. doi: 10.1038/ng.454. Epub 2009 Oct 4. PMID 19801981
- [Background] Schwab JH, Boland PJ, Agaram NP, Socci ND, Guo T, O'Toole GC, Wang X, Ostroumov E, Hunter CJ, Block JA, Doty S, Ferrone S, Healey JH, Antonescu CR. Chordoma and chondrosarcoma gene profile: implications for immunotherapy. Cancer Immunol Immunother. 2009 Mar;58(3):339-49. doi: 10.1007/s00262-008-0557-7. Epub 2008 Jul 19. PMID 18641983
- [Background] Oakley GJ, Fuhrer K, Seethala RR. Brachyury, SOX-9, and podoplanin, new markers in the skull base chordoma vs chondrosarcoma differential: a tissue microarray-based comparative analysis. Mod Pathol. 2008 Dec;21(12):1461-9. doi: 10.1038/modpathol.2008.144. Epub 2008 Sep 26. PMID 18820665
- [Background] Walcott BP, Nahed BV, Mohyeldin A, Coumans JV, Kahle KT, Ferreira MJ. Chordoma: current concepts, management, and future directions. Lancet Oncol. 2012 Feb;13(2):e69-76. doi: 10.1016/S1470-2045(11)70337-0. PMID 22300861
- [Background] Stacchiotti S, Sommer J; Chordoma Global Consensus Group. Building a global consensus approach to chordoma: a position paper from the medical and patient community. Lancet Oncol. 2015 Feb;16(2):e71-83. doi: 10.1016/S1470-2045(14)71190-8. PMID 25638683
- [Background] Dubory A, Missenard G, Lambert B, Court C. "En bloc" resection of sacral chordomas by combined anterior and posterior surgical approach: a monocentric retrospective review about 29 cases. Eur Spine J. 2014 Sep;23(9):1940-8. doi: 10.1007/s00586-014-3196-z. Epub 2014 Jan 28. PMID 24469886
- [Background] Asavamongkolkul A, Waikakul S. Wide resection of sacral chordoma via a posterior approach. Int Orthop. 2012 Mar;36(3):607-12. doi: 10.1007/s00264-011-1381-9. Epub 2011 Oct 29. PMID 22038441
- [Background] Stacchiotti S, Casali PG, Lo Vullo S, Mariani L, Palassini E, Mercuri M, Alberghini M, Pilotti S, Zanella L, Gronchi A, Picci P. Chordoma of the mobile spine and sacrum: a retrospective analysis of a series of patients surgically treated at two referral centers. Ann Surg Oncol. 2010 Jan;17(1):211-9. doi: 10.1245/s10434-009-0740-x. Epub 2009 Oct 22. PMID 19847568
- [Background] Varga PP, Szoverfi Z, Fisher CG, Boriani S, Gokaslan ZL, Dekutoski MB, Chou D, Quraishi NA, Reynolds JJ, Luzzati A, Williams R, Fehlings MG, Germscheid NM, Lazary A, Rhines LD. Surgical treatment of sacral chordoma: prognostic variables for local recurrence and overall survival. Eur Spine J. 2015 May;24(5):1092-101. doi: 10.1007/s00586-014-3728-6. Epub 2014 Dec 23. PMID 25533857
- [Background] Kayani B, Hanna SA, Sewell MD, Saifuddin A, Molloy S, Briggs TW. A review of the surgical management of sacral chordoma. Eur J Surg Oncol. 2014 Nov;40(11):1412-20. doi: 10.1016/j.ejso.2014.04.008. Epub 2014 Apr 25. PMID 24793103
- [Background] Puri A, Agarwal MG, Shah M, Srinivas CH, Shukla PJ, Shrikhande SV, Jambhekar NA. Decision making in primary sacral tumors. Spine J. 2009 May;9(5):396-403. doi: 10.1016/j.spinee.2008.10.001. Epub 2008 Dec 6. PMID 19059810
- [Background] Chen KW, Yang HL, Kandimalla Y, Liu JY, Wang GL. Review of current treatment of sacral chordoma. Orthop Surg. 2009 Aug;1(3):238-44. doi: 10.1111/j.1757-7861.2009.00027.x. PMID 22009849
- [Background] Gennari L, Azzarelli A, Quagliuolo V. A posterior approach for the excision of sacral chordoma. J Bone Joint Surg Br. 1987 Aug;69(4):565-8. doi: 10.1302/0301-620X.69B4.3611160.
- [Background] Clarke MJ, Dasenbrock H, Bydon A, Sciubba DM, McGirt MJ, Hsieh PC, Yassari R, Gokaslan ZL, Wolinsky JP. Posterior-only approach for en bloc sacrectomy: clinical outcomes in 36 consecutive patients. Neurosurgery. 2012 Aug;71(2):357-64; discussion 364. doi: 10.1227/NEU.0b013e31825d01d4. PMID 22569060
- [Background] Weitao Y, Qiqing C, Songtao G, Jiaqiang W. Use of gluteus maximus adipomuscular sliding flaps in the reconstruction of sacral defects after tumor resection. World J Surg Oncol. 2013 May 23;11:110. doi: 10.1186/1477-7819-11-110. PMID 23701700
- [Background] Doita M, Harada T, Iguchi T, Sumi M, Sha H, Yoshiya S, Kurosaka M. Total sacrectomy and reconstruction for sacral tumors. Spine (Phila Pa 1976). 2003 Aug 1;28(15):E296-301. doi: 10.1097/01.BRS.0000083230.12704.E3. PMID 12897508
- [Background] Zhang HY, Thongtrangan I, Balabhadra RS, Murovic JA, Kim DH. Surgical techniques for total sacrectomy and spinopelvic reconstruction. Neurosurg Focus. 2003 Aug 15;15(2):E5. doi: 10.3171/foc.2003.15.2.5. PMID 15350036
- [Background] Kim JE, Pang J, Christensen JM, Coon D, Zadnik PL, Wolinsky JP, Gokaslan ZL, Bydon A, Sciubba DM, Witham T, Redett RJ, Sacks JM. Soft-tissue reconstruction after total en bloc sacrectomy. J Neurosurg Spine. 2015 Jun;22(6):571-81. doi: 10.3171/2014.10.SPINE14114. Epub 2015 Mar 27. PMID 25815806
- [Background] Maricevich M, Maricevich R, Chim H, Moran SL, Rose PS, Mardini S. Reconstruction following partial and total sacrectomy defects: an analysis of outcomes and complications. J Plast Reconstr Aesthet Surg. 2014 Sep;67(9):1257-66. doi: 10.1016/j.bjps.2014.05.001. Epub 2014 May 20. PMID 24907194
- [Background] Imai R, Kamada T, Sugahara S, Tsuji H, Tsujii H. Carbon ion radiotherapy for sacral chordoma. Br J Radiol. 2011 Dec;84 Spec No 1(Spec Iss 1):S48-54. doi: 10.1259/bjr/13783281. Epub 2011 Mar 22. PMID 21427182
- [Background] Yanagi T, Kamada T, Tsuji H, Imai R, Serizawa I, Tsujii H. Dose-volume histogram and dose-surface histogram analysis for skin reactions to carbon ion radiotherapy for bone and soft tissue sarcoma. Radiother Oncol. 2010 Apr;95(1):60-5. doi: 10.1016/j.radonc.2009.08.041. Epub 2009 Sep 18. PMID 19767117
- [Background] Mima M, Demizu Y, Jin D, Hashimoto N, Takagi M, Terashima K, Fujii O, Niwa Y, Akagi T, Daimon T, Hishikawa Y, Abe M, Murakami M, Sasaki R, Fuwa N. Particle therapy using carbon ions or protons as a definitive therapy for patients with primary sacral chordoma. Br J Radiol. 2014 Jan;87(1033):20130512. doi: 10.1259/bjr.20130512. Epub 2013 Nov 28. PMID 24288399
- [Background] Uhl M, Edler L, Jensen AD, Habl G, Oelmann J, Roder F, Jackel O, Debus J, Herfarth K. Randomized phase II trial of hypofractionated proton versus carbon ion radiation therapy in patients with sacrococcygeal chordoma-the ISAC trial protocol. Radiat Oncol. 2014 Apr 29;9:100. doi: 10.1186/1748-717X-9-100. PMID 24774721
- [Background] Fossati P, Molinelli S, Matsufuji N, Ciocca M, Mirandola A, Mairani A, Mizoe J, Hasegawa A, Imai R, Kamada T, Orecchia R, Tsujii H. Dose prescription in carbon ion radiotherapy: a planning study to compare NIRS and LEM approaches with a clinically-oriented strategy. Phys Med Biol. 2012 Nov 21;57(22):7543-54. doi: 10.1088/0031-9155/57/22/7543. Epub 2012 Oct 26. PMID 23104051
- [Background] Steinstrater O, Grun R, Scholz U, Friedrich T, Durante M, Scholz M. Mapping of RBE-weighted doses between HIMAC- and LEM-Based treatment planning systems for carbon ion therapy. Int J Radiat Oncol Biol Phys. 2012 Nov 1;84(3):854-60. doi: 10.1016/j.ijrobp.2012.01.038. Epub 2012 Apr 6. PMID 22483698
- [Background] DeLaney TF, Liebsch NJ, Pedlow FX, Adams J, Dean S, Yeap BY, McManus P, Rosenberg AE, Nielsen GP, Harmon DC, Spiro IJ, Raskin KA, Suit HD, Yoon SS, Hornicek FJ. Phase II study of high-dose photon/proton radiotherapy in the management of spine sarcomas. Int J Radiat Oncol Biol Phys. 2009 Jul 1;74(3):732-9. doi: 10.1016/j.ijrobp.2008.08.058. Epub 2008 Dec 25. PMID 19095372
- [Background] DeLaney TF, Liebsch NJ, Pedlow FX, Adams J, Weyman EA, Yeap BY, Depauw N, Nielsen GP, Harmon DC, Yoon SS, Chen YL, Schwab JH, Hornicek FJ. Long-term results of Phase II study of high dose photon/proton radiotherapy in the management of spine chordomas, chondrosarcomas, and other sarcomas. J Surg Oncol. 2014 Aug;110(2):115-22. doi: 10.1002/jso.23617. Epub 2014 Apr 19. PMID 24752878
- [Background] Chen YL, Liebsch N, Kobayashi W, Goldberg S, Kirsch D, Calkins G, Childs S, Schwab J, Hornicek F, DeLaney T. Definitive high-dose photon/proton radiotherapy for unresected mobile spine and sacral chordomas. Spine (Phila Pa 1976). 2013 Jul 1;38(15):E930-6. doi: 10.1097/BRS.0b013e318296e7d7. PMID 23609202
- [Background] Staab A, Rutz HP, Ares C, Timmermann B, Schneider R, Bolsi A, Albertini F, Lomax A, Goitein G, Hug E. Spot-scanning-based proton therapy for extracranial chordoma. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):e489-96. doi: 10.1016/j.ijrobp.2011.02.018. Epub 2011 Apr 15. PMID 21497457
- [Background] Terezakis SA, Lovelock DM, Bilsky MH, Hunt MA, Zatcky J, Yamada Y. Image-guided intensity-modulated photon radiotherapy using multifractionated regimen to paraspinal chordomas and rare sarcomas. Int J Radiat Oncol Biol Phys. 2007 Dec 1;69(5):1502-8. doi: 10.1016/j.ijrobp.2007.05.019. Epub 2007 Aug 6. PMID 17689028
- [Background] Yamada Y, Laufer I, Cox BW, Lovelock DM, Maki RG, Zatcky JM, Boland PJ, Bilsky MH. Preliminary results of high-dose single-fraction radiotherapy for the management of chordomas of the spine and sacrum. Neurosurgery. 2013 Oct;73(4):673-80; discussion 680. doi: 10.1227/NEU.0000000000000083. PMID 23842548
- [Background] Zabel-du Bois A, Nikoghosyan A, Schwahofer A, Huber P, Schlegel W, Debus J, Milker-Zabel S. Intensity modulated radiotherapy in the management of sacral chordoma in primary versus recurrent disease. Radiother Oncol. 2010 Dec;97(3):408-12. doi: 10.1016/j.radonc.2010.10.008. Epub 2010 Nov 4. PMID 21056488
- [Background] Henderson FC, McCool K, Seigle J, Jean W, Harter W, Gagnon GJ. Treatment of chordomas with CyberKnife: georgetown university experience and treatment recommendations. Neurosurgery. 2009 Feb;64(2 Suppl):A44-53. doi: 10.1227/01.NEU.0000341166.09107.47. PMID 19165073
- [Background] Royston P, Parmar MK. The use of restricted mean survival time to estimate the treatment effect in randomized clinical trials when the proportional hazards assumption is in doubt. Stat Med. 2011 Aug 30;30(19):2409-21. doi: 10.1002/sim.4274. Epub 2011 May 25. PMID 21611958
- [Background] Stablein DM, Carter WH Jr, Novak JW. Analysis of survival data with nonproportional hazard functions. Control Clin Trials. 1981 Jun;2(2):149-59. doi: 10.1016/0197-2456(81)90005-2. PMID 7273792
- [Background] Li J, Scheike TH, Zhang MJ. Checking Fine and Gray subdistribution hazards model with cumulative sums of residuals. Lifetime Data Anal. 2015 Apr;21(2):197-217. doi: 10.1007/s10985-014-9313-9. Epub 2014 Nov 25. PMID 25421251
- [Background] McCandless LC, Gustafson P, Levy AR, Richardson S. Hierarchical priors for bias parameters in Bayesian sensitivity analysis for unmeasured confounding. Stat Med. 2012 Feb 20;31(4):383-96. doi: 10.1002/sim.4453. PMID 22253142
- [Background] Peduzzi P, Concato J, Feinstein AR, Holford TR. Importance of events per independent variable in proportional hazards regression analysis. II. Accuracy and precision of regression estimates. J Clin Epidemiol. 1995 Dec;48(12):1503-10. doi: 10.1016/0895-4356(95)00048-8. PMID 8543964
- [Background] Yuo TH, Degenholtz HS, Chaer RA, Kraemer KL, Makaroun MS. Effect of hospital-level variation in the use of carotid artery stenting versus carotid endarterectomy on perioperative stroke and death in asymptomatic patients. J Vasc Surg. 2013 Mar;57(3):627-34. doi: 10.1016/j.jvs.2012.09.036. Epub 2013 Jan 9. PMID 23312937